CLINICAL TRIAL: NCT03427138
Title: Investigating the Mirror Neuron System in Autism Spectrum Disorder
Brief Title: Training Early Social Language in Autism
Acronym: TESLA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Boston University Charles River Campus (Other)
Collaborators: University of Maryland, College Park (Other); University of Chicago (Other); Centre National de la Recherche Scientifique, France (Other); University of California, Los Angeles (Other); Boston Medical Center (Other)
Responsible Party: Principal Investigator, Helen B. Tager-Flusberg, Professor, Psychological & Brain Sciences, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4190E
Record Dates: First submitted 2018-01-23; First posted 2018-02-09 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Activator Appliances

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jasper (Experimental): JASPER (Joint Attention Symbolic Play Engagement Regulation) is a targeted intervention that focusses on early communication skills.
  Interventions: Behavioral: Jasper
- Parent Education (Experimental): Parent education intervention focusses on parenting a child with autism.
  Interventions: Behavioral: Parent Education

INTERVENTIONS:
Behavioral: Jasper — Families in the joint attention intervention will receive 10 weeks of the JASPER (Joint Attention Symbolic Play Engagement Regulation) protocol. JASPER is a treatment approach based on a combination of developmental and behavioral principles developed by Dr. Connie Kasari at the Center for Autism Research and Treatment, at University of California, Los Angeles. Our research staff will be trained on the specific techniques of JASPER guided by Connie Kasari (consultant on project) and her colleagues The study's intervention involves 2 days/week of 60-minute sessions with a trained experimenter (which may take place in the lab or home, depending on the needs of the family). The primary goal for the intervention will be to increase the frequency and range/variety of joint attention and to advance the child to higher levels (e.g., from requesting to initiating joint attention acts).
  Arms: Jasper
Behavioral: Parent Education — Families in the parent education intervention. Parent education will be provided in group sessions. During the sessions information is presented about ASD, how to deal with behavioral difficulties and available services, and parents are given an opportunity to share experiences. Parents will attend a weekly session for 10 weeks. 10 different topics will be discussed, which include: causes and symptoms of autism, diagnosis process, treatment options, enhancing communicative abilities in children with autism, emotion regulation, dealing with distress, correcting behavior difficulties, applying structure and routines.
  Arms: Parent Education

SUMMARY:
The aim of the study is to determine whether a targeted behavioral intervention can lead to both changes in early communication skills and in neural responses in toddlers and preschoolers with autism.

DETAILED DESCRIPTION:
The mirror neuron system (MNS) broadly refers to a network of brain regions that responds both when a person performs an action and when that person observes someone else performing the same action. This system emerges in infancy and develops over time to support more complex social abilities. It has been hypothesized that autism involves fundamental impairments to the MNS, which can explain the deficits in joint attention, imitation, communication and social cognition.

This study investigates the MNS in 100 toddlers and preschoolers recently diagnosed with autism or with a suspected diagnosis of autism. First, children with (suspected) autism complete a battery of behavioral measures and MNS activity will be assessed using electrophysiology (EEG; event-related potentials) while the child participates in specific tasks. Then, the children with (suspected) autism will be randomly assigned to one of two behavioral intervention programs (i.e., targeted joint attention intervention or parent education intervention) that will be carried out by interventionists and parents for 10-12 weeks. At the end of the intervention, these children will be re-evaluated on behavioral tasks and EEG to investigate changes as a result of the intervention.

The investigators hypothesize that the joint attention intervention will lead to significant changes on both the neural and behavioral measures of MNS functioning.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 18 and 59 months with a confirmed or suspected DSM5 diagnosis of autism spectrum disorder
* The included parents or guardians are required to be the primary caregivers of these children
* Families must speak English in the home at least 75% of the time.

Exclusion Criteria:

* Seizure disorder (may influence EEG data)
* Gestational age <32 weeks
* History of serious head trauma
* Genetic syndrome (e.g., fragile X syndrome)

Ages: 18 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in EEG Frequency Data- Resting State | Assessment occurs at week 1 and week 12, with an intervention in weeks 2-11
  EEG frequency data as measured during resting state
Change in EEG Frequency Data- Grasping Objects | Assessment occurs at week 1 and week 12, with an intervention in weeks 2-11
  EEG frequency data as measured while subjects grasps an object
Change in EEG Frequency Data- Observing actions | Assessment occurs at week 1 and week 12, with an intervention in weeks 2-11
  EEG frequency data as measured while child observes objects grasped and pointed to by others.
Change in joint attention measured with the Early Social and Communication scales (ESCS) | Assessment occurs at week 1 and week 12, with an intervention in weeks 2-11
  This behavioral assessment follows standardized guidelines to capture the full range of joint attention and behavior request skills (initiate and response). A child has a higher score on the ESCS when they demonstrate behavior requests (e.g. pointing to, or asking for, desired objects), or respond to behavior requests (e.g. giving objects to other people) and joint attention (e.g. three-point gaze). In the ESCS, a higher score would indicate higher social and communication abilities.
Change in play level measured with the Structured Play Assessment (SPA) | Assessment occurs at week 1 and week 12, with an intervention in weeks 2-11
  Developed by Ungerer & Sigman (1981), this assessment evaluates the child's number and variety of functional and symbolic play acts when introduced sequentially to 5 toy sets.
Change in imitation measured with the Elicited Imitation Battery (adapted from Rogers et al., 2003) | Assessment occurs at week 1 and week 12, with an intervention in weeks 2-11
  The child is presented with 3 manual actions (e.g., holding palm up), 3 actions on objects. The child's movements will be coded on a 5-point scale from 0 (no movement) to 5 (imitating all the different experimenter actions).
Change in language measured with the Elicitation of Language Sample Assessment-Toddler version (ELSA-T) | Assessment occurs at week 1 and week 12, with an intervention in weeks 2-11
  This 15-minute assessment is developed at the Center for Autism Research Excellence at Boston University. It evaluates expressive language abilities of participants.
Change in parent-child interactions | Assessment occurs at week 1, week 6, and week 12, with an intervention in weeks 2-11
  A 10-minute play-based parent-child interaction, using a standard set of age-appropriate toys will be recorded and used as part of the child's expressive language sample.
Change in predictive gaze measured with eye-tracking | Assessment occurs at week 1 and week 12, with an intervention in weeks 2-11
  During the EEG task, eye movements are recorded to assess the child's ability to predict action outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Tager-Flusberg, PhD, Principal Investigator — Boston University Charles River Campus
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
NDAR submission, including all measures
Supporting Information: Study Protocol
Time Frame: Currently available and continuing indefinitely
Access Criteria: By request through NDAR
URL: http://ndar.nih.gov

REFERENCES:
- See also: Lab webpage with information about the study — https://www.bu.edu/autism/participating-toddlers-with-autism/
- Available data/document: Individual Participant Data Set: C2495 — http://ndar.nih.gov